CLINICAL TRIAL: NCT05535023
Title: Phase 2 Study of Neoadjuvant SAR444245 Plus Cemiplimab in HPV Related Oropharynx
Brief Title: Phase 2 Study of Neoadjuvant SAR444245 Plus Cemiplimab in HPV Related Oropharynx Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0013; NCI-2022-07560 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-09-04; First posted 2022-09-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Squamous Cell Carcinoma; Oropharynx Cancer; Head and Neck Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Oropharyngeal Neoplasms; Head and Neck Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR444245 plus Cemiplimab (Experimental): Participants will receive SAR444245 and Cemiplimab by vein on Day 1 of Cycles 1 and 2. Each drug's infusion should take about 30 minutes.
  Interventions: Drug: SAR444245; Drug: Cemiplimab

INTERVENTIONS:
Drug: SAR444245 — Given by vein (IV)
Drug: Cemiplimab — Given by vein (IV)

SUMMARY:
To learn if SAR444245 given in combination with cemiplimab can help to kill cancer cells in patients with HPV-related oropharynx cancer who are scheduled to have surgery to remove the disease

DETAILED DESCRIPTION:
Primary Objective(s):

- To evaluate the major pathologic response (MPR; ≤ 10% residual tumor) rate of SAR444245 combined with cemiplimab administered in the neoadjuvant setting

Secondary Objective(s):

* To evaluate the safety and tolerability of neoadjuvant SAR444245 plus cemiplimab using NCI-CTCAE version 5.0
* To evaluate the feasibility of neoadjuvant SAR444245 plus cemiplimab by assessing the percentage of patients not able to undergo the initially proposed

surgery due to disease progression or an adverse event attributed to the drug combination

* To evaluate the objective response rate (ORR) to neoadjuvant SAR444245 plus cemiplimab by RECIST 1.1 (12)
* To evaluate the proportion of patients who changed TNM stage (ie: change of TNM stage post-treatment as compared to pre-treatment) followed neoadjuvant SAR444245 plus cemiplimab
* To assess the 1-year disease-free (DFS) survival rate

Exploratory Objective(s):

* To evaluate HPV cell-free DNA as a biomarker of response to therapy
* To evaluate pre- and post- treatment tumor and blood biomarkers and correlate with pathologic and clinical response and toxicity.
* To evaluate the relationship between matched time-point RECIST criteria on anatomic imaging (T1/T2 MRI or contrast CT) with candidate functional imaging (diffusion-weighted imaging, MR relaxometry, MRI/CT radiomics), pathologic (MPR) and serum (cfDNA) novel biomarkers of therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent and in this protocol
* Age ≥ 18 years old
* Newly diagnosed HPV-related oropharynx squamous cell carcinoma, either confirmed or suspected. Patients with a primary oropharynx cancer consistent with squamous cell carcinoma based on clinical presentation and radiological features AND that are interested in participating in this study can have histological confirmation at the same time as the research biopsy. Patient can only participate in the study if squamous cell carcinoma histology AND HPV is confirmed.
* Disease stage I per the TNM AJCC 8th Edition
* Patients must be amenable to TORS in the opinion of the treating head and neck surgeon
* Patients must be willing to undergo baseline biopsy to obtain tumor material
* Disease must be measurable by RECIST 1.1
* Performance status ECOG 0 or 1
* Baseline pulse oximetry > 92%
* Patients must have adequate normal organ and marrow function. Abnormal organ and marrow function is defined as:

neutrophils <1500/mm3, platelet count <100,000/mm3, hemoglobin <9 g/dL, total bilirubin >1.5 upper limit of normal (ULN) (except known Gilbert's syndrome), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.5 of upper limit of normality (ULN) Glomerular Filtration Rate (GFR) <40 mL/min/1.73 m2 (GFR will be calculated using the CKD-EPI equation per institutional standard)

- Female patients with reproductive potential must practice two effective contraceptive measures for the duration of study drug therapy and for at least 120 days after completion of study therapy. The two birth control methods can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom, copper intrauterine device, sponge,

or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).

* Male participants with female partners of childbearing potential are eligible to participate if they agree to either be abstinent from penile-vaginal intercourse or use a male condom plus partner use of a hormonal contraceptive method during the treatment period and for at least 120 days after the last dose of study treatment. Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration.
* Patient weight must be at least 50 Kg

Exclusion Criteria:

* History of previous malignancy other than malignancy treated with curative intent and with no evidence of active disease ≥3 years before the first dose of the study drugs and of low potential risk for recurrence. Patients with the following diagnoses represents an exception and may enroll:

  1. Non-melanoma skin cancers with no current evidence of disease
  2. Melanoma in situ with no current evidence of disease
  3. Localized cancer of the prostate with prostate-specific antigen of <1 ng/mL
  4. Treated or localized well-differentiated thyroid cancer
  5. Treated cervical carcinoma in situ
  6. Treated ductal/lobular carcinoma in situ of the breast
* International Normalized Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (aPTT) >1.5 × ULN unless the participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
* Participants under anti-hypertensive treatment who cannot temporarily (for at least 36 hours) withhold antihypertensive medications prior to each IMP dosing.
* Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti-fungal therapy ≤14 days prior to administration of investigational product. Patients with known hepatitis B, hepatitis C (HCV), or HIV infection could go on study provided the viral load is undetectable at Screening.
* Unstable or severe uncontrolled medical condition (e.g., unstable cardiac or pulmonary function or uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the risk to the patient associated with his or her participation in the study.
* Female subjects who are pregnant or breast-feeding
* Known hypersensitivity (≥ Grade 3) to or contraindication for the use of any study intervention or components thereof, including premedication to be administered in this study, as well as PEG or any pegylated drug and E. coli-derived protein".
* Patient with active, known, or suspected autoimmune disease that has required systemic therapy. Exceptions: patients with vitiligo, type I diabetes mellitus, and endocrinopathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | through study completion an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org